CLINICAL TRIAL: NCT04242433
Title: Patterns of Resistance-associated Substitutions in Patients With Chronic HCV Infection Following Treatment With Direct Acting Antiviral Agents in the Public Health Setting
Brief Title: HCV RAS Testing in Public Health Programs
Acronym: RAS-HCV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Radha K Dhiman, Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: IEC-2018-867
Record Dates: First submitted 2019-10-07; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Hepatitis C; Public Health; Direct Acting Antiviral Agents; Resistance Associated Substitutions
Keywords: Resistance associated substitutions; HCV
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum will be stored with HCV RNA samples in the institutions's secure facility
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Viremic Person living with HCV: All persons enrolled in the MMPHCRF treatment programme are provided free of charge direct acting antiviral agents and followed up for outcomes.
  Interventions: Drug: Direct Acting Antivirals

INTERVENTIONS:
Drug: Direct Acting Antivirals — All subjects with viremic chronic hepatitis C will be given DAAs based on the MMPHCRF Treatment algorithm. Patients will be assessed for cirrhosis, prior treatment exposure, high risk groups like dialysis patients, HIV-HCV coinfection, etc. Accordingly treatment will be provided at any of the 25 peripheral centres or at the apex nodal treatment centre (PGIMER) of the MMPHCRF.
  Baseline and post treatment RAS samples will be collected with consent.

SUMMARY:
Successful treatment of hepatitis C has been reported to be associated with 62-84% reduction in all-cause mortality (deaths), 68-79% reduction in risk of HCC and 90% reduction in risk of liver transplantation. The efficacy of NS5A inhibitors for the treatment of patients chronically infected with hepatitis C virus (HCV) can be affected by the presence of NS5A resistance-associated substitutions (RASs). Pre-existence of resistance associated substitutions (RASs) to direct antiviral agents (DAAs) reduces sustained virologic response (SVR) rates by 3-53% in hepatitis C virus (HCV) genotype 3 infected patients depending on different predictors and the DAA regimen used. This study will prospectively analyze data from the MukhMantri Punjab Hepatitis C Relief Fund (MMPHCRF) to determine the posttreatment prevalence of various NS5A RASs, and their effect on outcomes of treatment with daclatasvir-sofosbuvir or sofosbuvir-ledipasvirin patients with chronic HCV.

The study aims to assess the prevalence and effect of RASs on sustained virological response (SVR) rates in patients with treatment failure to a regimen containing sofosbuvir and ledipasvir/daclatasvir.

ELIGIBILITY:
Inclusion Criteria:

* All viremic chronic hepatitis C

Exclusion Criteria:

* People with disseminated malignancy, advanced cardiovascular, 18 pulmonary, or neurological disease with short life expectancy were not enrolled

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The MMPHCRF Cohort patients are treated at 25 sites in Punjab State India with algorithm based DAAs for chronic Hepatitis C.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-07-16 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Achievement of sustained virological response | 12 weeks after treatment completion
  SVR12
Assessment of RAS | 12 weeks after treatment completion
  12 weeks after treatment completion

SECONDARY OUTCOMES:
Assessment of RAS in treatment failures | 12 weeks after treatment completion
  Comparison of variants in those who achieve or fail to achieve SVR12

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - Postgraduate Institute of Medical Education and Research, Chandigarh

IPD SHARING:
Plan to Share IPD: Undecided